CLINICAL TRIAL: NCT04583553
Title: Comparative Microbial Analysis of Cystitis in Non-muscle-invasive Bladder Cancer Patients Using Vikor Scientific Urine-IDTM and Standard Laboratory Culture
Brief Title: Comparative Microbial Analysis of Cystitis in Non-muscle-invasive Bladder Cancer Patients Using Vikor Scientific Urine-ID Testing Menu (IDTM) and Standard Laboratory Culture
Acronym: VS-UrineID
Status: Withdrawn | Type: Observational
Why Stopped: Site did not proceed with study.
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Vikor Scientific (Unknown)
Responsible Party: Principal Investigator, Eugene Lee, MD, Associate Professor, University of Kansas Medical Center
Other Study IDs: VS-UrineID
Record Dates: First submitted 2020-10-05; First posted 2020-10-12 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Urinary Tract Infections; Bladder Cancer
MeSH Terms: conditions — Urinary Tract Infections; Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine Samples will be collected for study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Vikor Scientific Urine-IDTM — Urine samples will be collected for both standard laboratory culture at KUMC Lab and expedited delivery to Vikor Scientific Lab for Urine-IDTM analysis. Vikor Scientific will cover all costs associated with sample delivery. If insufficient urine volume is collected for both standard laboratory culture at KUMC Lab and Vikor Scientific Urine-IDTM, urine will be preferentially used for standard laboratory culture at KUMC Lab.

SUMMARY:
Vikor Scientific Urine-IDTM is a molecular analysis technology which provides pathogen detection, quantification, and resistance gene identification. Urine-IDTM delivers its results through the technology platform Antibiotic Stewardship program (ABXAssist™), which provides results incorporating regional sensitivity and susceptibility patterns, medication costs, antibiotic spectrum of activity, and FDA guidance. This product aims to deliver prompt, patient-centered and value-based guidance to clinicians for antibiotic selection within 24 hours of delivery to testing facility.

Proposed advantages of Vikor Scientific Urine-IDTM include:

* Expeditious result (within 24 hours post-lab arrival)
* Simultaneous detection of polymicrobial and monomicrobial infections
* Identification of 49 most common antibiotic resistance genes
* Provision of up-to-date regional sensitivity and susceptibility patterns
* Provision of cost-sensitive treatment options and FDA guidance
* Easy accessibility (mobile, web-portal and electronic health records Integration)

This utility of this technology has yet to be investigated in a clinical study and could prove to be a viable alternative or adjunctive diagnostic tool to standard laboratory culture. Standard laboratory culture can take up to 7 days to return pathogen identification and antibiotic susceptibility, potentially delaying appropriate care and prolonging exposure to inappropriate empiric antibiotics. Our study aims to analyze the ability Vikor Scientific Urine-IDTM to improve time to identification of correct pathogen and accuracy of pathogen identification when compared to standard laboratory culture.

DETAILED DESCRIPTION:
Commercially available Vikor Scientific Urine-IDTM urine collection kits will be provided to the University of Kansas Medical Center (KUMC) Department of Urology by Vikor Scientific.

Urine samples will be collected for both standard laboratory culture at KUMC Lab and expedited delivery to Vikor Scientific Lab for Urine-IDTM analysis. Vikor Scientific will cover all costs associated with sample delivery. If insufficient urine volume is collected for both standard laboratory culture at KUMC Lab and Vikor Scientific Urine-IDTM, urine will be preferentially used for standard laboratory culture at KUMC Lab.

Provider clinical decision making will be based on standard laboratory cultures and therapy will not be adjusted based on Vikor Urine-IDTM results.

ELIGIBILITY:
Inclusion Criteria:

1. Ability of participant OR Legally Authorized Representative (LAR) to understand this study, and participant or LAR willingness to provide informed consent.
2. Age ≥ 18 years
3. Diagnosis of Non-Muscle Invasive Bladder Cancer (NMIBC)
4. Onset of cystitis or UTI symptoms within 7 days of Transurethral Resection of the Bladder Tumor (TURBT) or BCG installation
5. Ability to collect urine sample for analysis via standard laboratory culture and Vikor Scientific Urine-IDTM

Exclusion Criteria:

1. Inability of participant OR Legally Authorized Representative (LAR) to understand this study, and participant or LAR willingness provide informed consent
2. Age <18 years
3. Diagnosis of Muscle-Invasive or metastatic bladder cancer
4. Onset of cystitis greater than 7 days following TURBT or BCG installation
5. Inability to provide sufficient urine for both standard laboratory culture and Vikor Scientific Urine-IDTM
6. Current prophylactic antibiotic use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All study participants will be enrolled from KUMC hospital and clinics. A total of 175 participants will be recruited. Participants undergoing the study will be asked to submit urine sample to KUMC Lab within 7 days of onset on cystitis symptoms. Urine sample will be divided for use in standard laboratory culture and Vikor Scientific Urine-IDTM. Urine-IDTM samples will be collected with kits provide by Vikor Scientific. Urine-IDTM kits will be expedited to Vikor Scientific Lab immediately following collection.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-12-15 (Estimated); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
To determine if Vikor Scientific Urine-IDTM can identify pathogen (or absence thereof) causing post-TURBT or post-bacillus Calmette Guerin (BCG) cystitis in a timelier manner than standard laboratory culture. | 2 years
To determine if Vikor Scientific Urine-IDTM provides concordant identification or urinary pathogen and antimicrobial sensitivity compared to standard laboratory culture in post-TURBT or post-BCG cystitis. | 2 years

SECONDARY OUTCOMES:
To characterize the pathogens involved in post-TURBT and post-BCG Urinary Tract Infection (UTI) and their antibiotic susceptibility/resistance profile | 2 years
To determine the prevalence of post-TURBT and post-BCG cystitis with no causative pathogenic organism | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Lee, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medcial Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No
Data will be analyzed at KUMC and published